Official Title: The Effect of Symptom Management Training Given to Gynaecological Cancer Patients Receiving Chemotherapy with Artificial Intelligence Supported Mobile Application on Supportive Care Needs, Symptom Severity and Psychological Well-Being

NCT number: NCT ID not yet assigned

ID: 2024-442

**Document Date:10.09.2024** 

## Statistical Analysis Plan

## **G-POWER ANALYSIS**



The study will be conducted with a total of 70 patients, including 35 patients from the intervention group and 35 patients from the control group (The sample number of the study was calculated by using the G Power programme using the data of a study in which mobile application intervention was carried out on cancer patients. Accordingly, the confidence interval was 95%; the margin of error was accepted as 5% and a total of 56 patients were found as 28 intervention and 28 control group. Considering that there may be losses during the mobile application intervention, the sample number was kept 25% higher than the calculated sample number.)

## Statistical Analysis

Statistical Package for Social Science (SPSS) 24.0 package programme will be used for statistical analysis of the data.

Data related to the descriptive and clinical characteristics of the participants will be evaluated by number, percentage, mean and standard deviation.

The similarities of the intervention and control groups in terms of descriptive and clinical characteristics will be evaluated.

Chi-square test for categorical variables and Mann Whitney U test for numerical variables will be used to determine whether the groups are similar in terms of some characteristics.

| The conformity of the scale scores to normal distribution will be evaluated by Shapiro-Vest. | VV IIK |
|---|---|